CLINICAL TRIAL: NCT06397469
Title: Optimizing a Closed-loop Digital Meditation Intervention for Remediating Cognitive Decline and Reducing Stress in Older Adults
Brief Title: Enhancing Attention and Wellbeing Using Digital Therapeutics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AG076668; 5R01AG076668 (NIH)
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Aging; MCI; Cognitive Decline
Keywords: healthy aging; attention; cognition; dementia; intervention; digital; behavioral; prevention; decline; stress reduction; Quality of life
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- MediTrain 30m/day for 6wks (Experimental): Participants will engage with a digital meditation app for the time listed above.
  Interventions: Device: MediTrain
- MediTrain 15m/day for 6wks (Experimental): Participants will engage with a digital meditation app for the time listed above.
  Interventions: Device: MediTrain
- MediTrain 30m/day for 3wks (Experimental): Participants will engage with a digital meditation app for the time listed above.
  Interventions: Device: MediTrain
- MediTrain 15m/day for 3wks (Experimental): Participants will engage with a digital meditation app for the time listed above.
  Interventions: Device: MediTrain
- Active Control Group (Active Comparator): An active control application will be used for this arm. The total training experience here will be for 6 weeks (5 days/week), with each training session lasting ~30 minutes (not including self-paced breaks). Here an app that is matched in terms of expectancy of benefits compared to our training groups will be determined by questioning 100 naïve individuals to predict their expected improvement on each cognitive domain across a multitude of possible applications.
  Interventions: Device: Worder

INTERVENTIONS:
Device: MediTrain — MediTrain is a tablet-based, meditation-inspired, cognitive training game aimed at improving self-regulation of internal attention and distractions. It was developed in collaboration with meditation thought-leader Jack Kornfield, and Zynga, a world-class video game company. It was created to make benefits of concentrative meditation more easily accessible to anyone, including complete novices. This is achieved by creating a game that yields quantifiable and attainable goals, provides feedback, and includes an adaptive algorithm to gradually increase difficulty as users improve.
  Arms: MediTrain 15m/day for 3wks; MediTrain 15m/day for 6wks; MediTrain 30m/day for 3wks; MediTrain 30m/day for 6wks
Device: Worder — Worder was designed to enhance visual motor and visual spatial skills in individuals of all ages and cognitive abilities. Visual processing is required for all cognitive abilities that involve vision including attention, working memory, and task management. Worder's goal is to improve cognitive function more broadly by developing this critical skill underlying multiple abilities.
  Arms: Active Control Group

SUMMARY:
The goals of the proposed research are to first determine the minimal and/or optimal dose of a digital intervention required for cognitive enhancement, and then to examine the impact of several potential moderators of treatment effects (i.e., cognitive decline, AD polygenic hazard score, cardiovascular risk, and race/ethnicity). This knowledge gained from his high-impact study with transform the field of cognitive interventions, paving the way for a precision medicine model for cognitive enhancing interventions that improve quality of life for older adults and individuals with cognitive deficits at risk of developing dementia.

ELIGIBILITY:
Inclusion Criteria:

* 60+ years old (adult)
* English language fluency
* owning a smartphone or tablet

Exclusion Criteria:

* Under 60 years old (minor)

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change on the Mobile Continuous Performance Task (CPT) over time | baseline, immediate follow-up, and at a 6 month follow-up
  The CPT is a 23-minute task, where participants are instructed to respond to target stimuli (squares at the top of the screen) and withhold responses to non-target stimuli (squares at the bottom of the screen). Performance will be quantified as: (1) mean reaction times, (2) standard deviation of reaction times (RTV), and (3) d-prime (comparing correct target detections or 'hits' to incorrect non-target detections or 'false alarms').

SECONDARY OUTCOMES:
Change on the Adaptive Cognitive Evaluation (ACE) over time | baseline, immediate follow-up, and at a 6 month follow-up
  The ACE is a mobile cognitive assessment tool, which includes a battery of cognitive control tests for rapid tests of cognition. The sub-tests (or 'modules') in ACE are adapted from standardized tasks to rapidly assess various aspects of cognition, including attention, memory, and multitasking. We will assess response time, accuracy, and response time variability in each case, with faster/more accurate/less variable performance being indicative of improved cognitive control.

OTHER OUTCOMES:
Mean Change on Everyday Cognition Scale (ECog) | baseline, immediate follow-up, and at a 6 month follow-up
  • Mean Change on Everyday Cognition Scale (ECog) The Everyday Cognition Scale (ECog) measures the ability to perform everyday tasks that demand memory, language, visuospatial abilities, planning, organization, and divided attention. The ECog consists of a global and domain scores for each of the previously described categories, and is scored as follows: 1= better or no change compared to 10 years earlier, 2= questionable/occasionally worse compared to 10 years earlier, 3= consistently a little worse compared to 10 years earlier, 4= consistently much worse compared to 10 years earlier. Thus, the lower the overall score is on this measure at both the global and domain score level, the better one is performing with respect to their cognition.
Mean Change on Pittsburgh Sleep Quality Index (sleep) | baseline, immediate follow-up, and at a 6 month follow-up
  • Pittsburgh Sleep Quality Index (sleep) The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Overall scores range from 0 to 21, with lower scores representing healthier sleep quality. We will report change in means over time.
Mean Change on Framingham Cardiovascular Risk Score | baseline, immediate follow-up, and at a 6 month follow-up
  • Framingham Cardiovascular Risk Score The Framingham Risk Score is a sex-specific algorithm used to estimate the 10-year cardiovascular risk of an individual. We will use the BMI version of the score. Scores range from 0-100% risk of cardiac event or death. We will report change in means over time.
Mean Change on SF-36 (overall health) | baseline, immediate follow-up, and at a 6 month follow-up
  • SF-36 (overall health) The general health and well-being (SF-36) score assesses participant health. The SF-36 score ranges from 0 to 100. The higher the overall score is on this measure, the better one is performing with respect to their health and well-being.
Mean Change on Cognitive Failures Questionnaire | baseline, immediate follow-up, and at a 6 month follow-up
  • Cognitive Failures Questionnaire (Distractibility) The Cognitive Failures Questionnaire (CFQ) assesses participant distractibility. The CFQ score ranges from 0 to 100, with the lower the overall score is on this measure, the better one is performing with respect to their cognition.
Mean Change on Perceived Stress Scale | baseline, immediate follow-up, and at a 6 month follow-up
  • Perceived Stress Scale A survey that measures the degree to which situations in one's life are perceived as stressful. Scores range from 0 to 40 with higher scores representing more perceived stress. We will report change in means over time.
Mean Change on UCLA 3-item Loneliness Scale | baseline, immediate follow-up, and at a 6 month follow-up
  * UCLA 3-item Loneliness Scale This is a very short 3-item measure that assesses how often a person feels disconnected from others. Scores range from 0-3 with 3 representing more loneliness. We will report change in means over time.
Mean Change on GAD-7 (anxiety) | baseline, immediate follow-up, and at a 6 month follow-up
  • GAD-7 (anxiety) The GAD-7 is a 7-item screening tool for generalized anxiety disorder. GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety. We will report change in means over time.
Mean Change on PHQ-9 (depression) | baseline, immediate follow-up, and at a 6 month follow-up
  • PHQ-9 (depression) The PHQ-9 is a 9-item scale that objectifies the degrees of depression severity a person is experiencing. Scores range from 0-27 with higher scores representing more depression. Scores at or below 4 suggest minimal or no depression. We will report change in means over time.
Mean Change on Emotional Regulation Questionnaire | baseline, immediate follow-up, and at a 6 month follow-up
  • Emotional Regulation Questionnaire A survey assessing a person's ability to manage and respond to emotional experiences. Scores range from 6 to 42 with higher scores representing more positive emotions. We will report change in means over time.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Gazzaley, MD/PhD, Principal Investigator — University of California, San Francisco; David Ziegler, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No